CLINICAL TRIAL: NCT02477137
Title: PhONEME - PartipatOn Ehealth MobilE. Effects of an Interactive Information and Communications Technology (ICT) Platform for Assessment and Management of Symptoms in Patients Treated for Prostate Cancer
Brief Title: Effects of an Interactive ICT-Platform for Assessment and Management of Symptoms in Patients Treated for Prostate Cancer
Acronym: PhONEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ann Langius-Eklöf, PhD, RN, Professor, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PhONEME Prostate
Record Dates: First submitted 2015-06-12; First posted 2015-06-22 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Nursing; Health Literacy; Quality of Life; Radiotherapy; Oncology Nursing; Self Care; Symptom Management; Participatory Care; Person-centered Care; Information and Communication Technology; Patient-reported symptoms; Mobile device
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): In combination with usual care according to the routines at the clinic, patients in the intervention group are given access to an application for a smartphone/tablet for daily reporting of symptoms, access to self-care advice and health-care professionals in real time.
  Interventions: Device: smartphone or tablet
- Control group (No Intervention): Usual care according to the routines at the clinic.

INTERVENTIONS:
Device: smartphone or tablet — Patients in the intervention group are given access to an application for a smartphone/tablet for daily reporting of symptoms, access to self-care advice and health-care professionals in real time.
  Other Names: Intervention
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate the effects of an interactive ICT-platform for use in a smartphone or tablet in patients treated with radiotherapy for prostate cancer. The hypothesis is that clinical management will be improved and costs reduced and safe and participatory care promoted, when patients report symptoms in an application which provides self-care advice and instant access to professionals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate cancer without metastases or spread to the lymph nodes,
* will receive radiation therapy for at least five (5) weeks,
* literacy in the Swedish language

Exclusion Criteria:

* Patients who need an interpreter at the doctor's visit
* Patients who have a known severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Questionnaire Scale for Functional Health Literacy (S-FHL - Swedish version) | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of understanding and communicating health
Questionnaire Individualized Care Scale (ICS) | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of individualized care as measured by the ICS
Questionnaire Sense of Coherence Scale (KASAM) | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of Sense of Coherence
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of health related quality of life
EORTC Prostate-specific module (QLQ-PR25) Questionnaire | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of symptom prevalence, characteristics and distress related to prostate cancer
Scale for Communicative and Critical Health Literacy (S-C & C HL - Swedish version) | up to 3 months after completion of radiotherapy treatment
  To evaluate self-reported data in terms of health literacy

SECONDARY OUTCOMES:
Health care costs | up to 3 months after completion of radiotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ann Langius-Eklöf, RN, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Crafoord MT, Ekstrand J, Sundberg K, Nilsson MI, Fjell M, Langius-Eklof A. Mobile Electronic Patient-Reported Outcomes and Interactive Support During Breast and Prostate Cancer Treatment: Health Economic Evaluation From Two Randomized Controlled Trials. JMIR Cancer. 2025 Mar 11;11:e53539. doi: 10.2196/53539. PMID 40067346
- [Derived] Langius-Eklof A, Crafoord MT, Christiansen M, Fjell M, Sundberg K. Effects of an interactive mHealth innovation for early detection of patient-reported symptom distress with focus on participatory care: protocol for a study based on prospective, randomised, controlled trials in patients with prostate and breast cancer. BMC Cancer. 2017 Jul 4;17(1):466. doi: 10.1186/s12885-017-3450-y. PMID 28676102